CLINICAL TRIAL: NCT04914533
Title: Exploratory Real-world Study Examining the Effect of the Luminance RED Device on Recurrent Aphthous Ulcer Stomatitis
Brief Title: Luminance RED for Canker Sores
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: did not launch
Sponsor: ProofPilot (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2795
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Canker Sore
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Intervention Model Description: Single arm trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention Arm (Experimental): Luminance Red Treatment Arm
  Interventions: Device: Luminance RED Low Level Laser Therapy Device

INTERVENTIONS:
Device: Luminance RED Low Level Laser Therapy Device — Low Level Laser Therapy (LLLT) sometimes known as Low Level Light Therapy or Photobiomodulation (PBM) is a low-intensity light therapy. The effect is photochemical not thermal. The Luminance RED Device is specifically designed to make it easy to issue LLLT to canker sores.

SUMMARY:
Canker sores, also called aphthous ulcers, are small, shallow lesions that develop on the soft tissues in your mouth or at the base of your gums. Unlike cold sores, canker sores don't occur on the surface of your lips and they aren't contagious. They can be painful, however, and can make eating and talking difficult. Recurrent aphthous ulcer stomatitis (RAS) is characterized by recurrent bouts of solitary or multiple shallow painful ulcers, at intervals of a few months to a few days in patients who are otherwise well.

Low Level Laser Therapy (LLLT) sometimes known as Low Level Light Therapy or Photobiomodulation (PBM) is a low-intensity light therapy. The effect is photochemical not thermal. The light triggers biochemical changes within cells and can be compared to the process of photosynthesis in plants, where the photons are absorbed by cellular photoreceptors, which trigger chemical changes.

The main medical usage of LLLT is for pain and inflammation reduction, promoting the regeneration of different tissues and preventing damage to tissues. With the use of the appropriate power (from 5 to 200mW) and wavelength (600-900nm), the therapy brings anti-inflammatory and analgesic results aiding in wound healing. The mechanism of action of LLLT may be very beneficial in the treatment of oral erosions and ulcers, however, very few studies have been performed on the treatment of RAS with LLLT. There are few reports on accelerated healing in erosive mucocutaneous disorders and they are often presented as a case series rather than large randomized clinical trials. The effects on skin wound healing and periodontal inflammation management with laser biostimulation suggest that this treatment modality may also be useful for oral erosive conditions.

This clinical trial aims to evaluate the effect of the Luminance RED device on the management of RAS.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* 18 years and older.
* Self report canker sore outbreaks once every 30 days or more frequent
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* No previous experience of LLLT.
* United States resident.
* Willingness and ability to submit a $49 deposit using a credit card for the device.

Exclusion Criteria:

* Patients with a known systemic disease that predisposes them to RAS (e.g., Behçet disease) or undergoing systemic treatment for RAS.
* The presence of a serious medical condition.
* Currently known to be pregnant or breastfeeding
* Patients treated with topical or systemic medication for RAS, such as corticosteroid therapy, antibiotics or analgesics during the previous month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-21 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-28 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Pain Scale | Baseline to day 18
  daily score of canker sore pain
Change in Eating, drinking, and brushing teeth questionnaire | Baseline to day 18
  score calculated on daily discomfort with eating, drinking and brushing teath

SECONDARY OUTCOMES:
Device retention | Day 21
  Percentage of participants who decide to keep device

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Amsden, Principal Investigator — ProofPilot
Locations (1):
- ProofPilot Virtual Online Trial (https://proofpilot.com), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided